CLINICAL TRIAL: NCT05417113
Title: Evaluation of the Addition of Liposomal Bupivacaine to the Erector Spinae Plane (ESP) Block to Multilevel Lumbar Spinal Fusion Surgery
Brief Title: Erector Spinae Block for Spine Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Christina Jeng, MD, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-22-00168
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine only (Active Comparator): bupivacaine 0.25% in ESP blocks
  Interventions: Drug: Bupivacaine
- Liposomal Bupivacaine and Bupivacaine (Experimental): liposomal bupivacaine in addition to 0.25% bupivacaine in ESP blocks
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — liposomal bupivacaine
  Arms: Liposomal Bupivacaine and Bupivacaine
Drug: Bupivacaine — bupivacaine 0.25% in ESP blocks

SUMMARY:
This study is to determine whether or not the addition of liposomal bupivacaine in an ESP block will have long term benefits for patients undergoing lumbar spinal fusion surgery. Given previous studies found long term benefits from liposomal bupivacaine, the hypothesis is that patients will have decreased opioid usage and improved pain scores when compared to a standard ESP block with plain 0.25% bupivacaine.

DETAILED DESCRIPTION:
This will be a double blind prospective randomized control trial comparing liposomal bupivacaine with plain bupivacaine in their effectiveness in ESP blocks in lumbar spinal fusion surgery. Patients scheduled for a lumbar spinal fusion procedure will be identified at the time of the scheduled surgery. The endpoints of this study include:

The primary objective is to compare the amount of postoperative intravenous opioid consumption among two study groups for the first 72 hours: Patients undergoing posterior lumbar spinal fusion surgery (1-2 levels) under general anesthesia and ESP block with liposomal bupivacaine + 0.25% bupivacaine and patients undergoing posterior lumbar spinal fusion surgery (1-2 levels) under general anesthesia and ESP block with 0.25% bupivacaine

The secondary objectives include:

Compare the severity of pain at rest at specific timepoints postoperatively. Compare general quality of recovery via QoR-15 at 48 hours, 72 hours and then at routine follow up visits occurring 2 weeks, 6 weeks, and 12 weeks postoperatively.

Measure rate of postoperative nausea/vomiting in PACU. Measure time to ambulation. Compare analgesia satisfaction score at time of discharge. Measure hospital length of stay.

ELIGIBILITY:
Inclusion criteria:

* Adults aged greater than or equal to 18 years old and less than or equal to 85 years old.
* Patients who are scheduled to undergo lumbar spinal surgery (1-2 level) and willing and able to provide informed consent.

Exclusion criteria:

* Patients with a history of chronic opioid use for > 3 months including but not limited to fentanyl, morphine, oxycodone, methadone.
* Patients with known allergy or intolerance to any drug used in the study including local anesthetics and total intravenous anesthesia medications.
* Patients with a history of alcohol or drug abuse.
* Patients with a history of intolerance of nonsteroidal anti-inflammatory drugs.-Patients with hepatic insufficiency.
* Patients with renal insufficiency.
* Patients who are pregnant.
* Patients with American Society of Anesthesiologists physical status of 4 or greater.
* Patients on immunosuppressive therapy. Pregnant patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jeng, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IRB approval was not obtained to share IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Started | 7 | 6
Completed | 5 | 4
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (13.35) | 63.3 (6.70) | 63.44 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 80.58 (17.23) | 78.88 (22.49) | 79.82 (18.41)
ASA Physical Status [Mean (Standard Deviation); unit: units on a scale] — ASA I A normal healthy patient
  ASA II A patient with mild systemic disease
  ASA III A patient with severe systemic disease
  ASA IV A patient with severe systemic disease that is a constant threat to life
  ASA V A moribund patient who is not expected to survive without the operation
  ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2.2 (0.45) | 2.5 (0.58) | 2.33 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Consumption During First 72 Hours
Description: The amount of postoperative intravenous opioid consumption (Total morphine mg equivalents MME) during the first 72 hours
Time Frame: 12 hours, 24 hours, 48 hours, 72 hours
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 5 | 4
MME
  12 hours | 11.69 (8.26) | 22.63 (4.02)
  24 hours | 19.56 (13.14) | 39.79 (19.36)
  48 hours | 30.66 (32.46) | 73.88 (15.05)
  72 hours | 38.99 (39.03) | 93.42 (31.35)

2. Secondary Outcome: Change in Pain Score
Description: Change in the severity of pain at rest using an 11-point Likert scale. Scale from 0-10, with higher score indicating more pain.
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 5 | 4
score on a scale
  1 hour post-operatively | 4.0 (2.74) | 4.5 (3.11)
  6 hours post-operatively | 2.0 (1.41) | 4.5 (3.87)
  12 hours post-operatively | 2.6 (4.34) | 3.75 (3.30)
  24 hours post-operatively | 2.8 (2.77) | 5.5 (2.89)
  48 hours post-operatively | 5.6 (3.78) | 5.0 (3.56)
  72 hours post-operatively | 5.0 (3.61) | 5.0 (3.56)
  2 weeks hours post-operatively | 4.6 (2.30) | 4.25 (2.06)
  6 weeks hours post-operatively | 2.4 (3.36) | 3.75 (4.19)
  12 weeks hours post-operatively | 2.2 (3.19) | 3.0 (1.41)

3. Secondary Outcome: Quality of Recovery (QOR 15)
Description: Change in general quality of recovery using a 15 point questionnaire via QoR-15 with regard to how the patient is feeling scored on a scale from 0-10, with 0 being none of the time and 10 being all of the time. Full scale range from 0-150, with a higher score indicating a better health outcome.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 5 | 4
score on a scale | 123.2 (7.39) | 108.0 (35.15)

4. Secondary Outcome: Number of Participants With Postoperative Nausea/Vomiting (PONV)
Description: Number of participants with postoperative nausea/vomiting (PONV) in PACU
Time Frame: in PACU (4 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

5. Secondary Outcome: Time to Ambulation
Description: Time to ambulation in hours
Time Frame: average 26-27 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 5 | 4
hours | 26.03 (12.58) | 27.13 (14.94)

6. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay (LOS)
Time Frame: average 72 hours
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 5 | 4
days | 3 (2.35) | 3.5 (0.58)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine and Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
Very limited enrollment due to volume of relevant surgeries and patient eligibility. Opioid consumption confounded by nonuniform usage of PCAs post-operatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT05417113/Prot_000.pdf
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT05417113/ICF_001.pdf